CLINICAL TRIAL: NCT03771612
Title: Inflammation and Daily Life Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Naomi Eisenberger, Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IDL; 1R21AG058893-01A1 (NIH)
Record Dates: First submitted 2018-12-06; First posted 2018-12-11 (Actual); Results first posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Inflammation
Keywords: Immune system; Social psychology; Health psychology
MeSH Terms: conditions — Inflammation | interventions — Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Naproxen (Active Comparator)
  Interventions: Drug: Naproxen
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Naproxen — Half of the participants will be randomly assigned to receive naproxen twice daily (400 mg total daily; 200 mg 2x a day)
  Arms: Naproxen
Drug: Placebos — Half of the participants will be randomly assigned to receive a placebo pill twice daily
  Arms: Placebo

SUMMARY:
UCLA researchers looking for healthy individuals (age 45-60) to participate in a study investigating whether an anti-inflammatory medication can impact daily life experiences.

Everyday for two weeks, participants will take either an anti-inflammatory medication (naproxen) twice daily, or a placebo pill twice daily. Participants will also answer daily questions during the 2-week period. Participants will also fill out questionnaires and complete a few tasks on the computer: once prior to the 2-week period and once immediately after the 2-week period, both during online study sessions.

DETAILED DESCRIPTION:
Participants (ntotal=50) will be men and women, ages 45-60. All interested participants will first complete a structured telephone interview in order to assess eligibility.

The study will begin with filling out questionnaires, as well as an online session to complete some tasks. You will then be randomly assigned to take either an anti-inflammatory medication (naproxen) or placebo (inactive substance) to take twice daily everyday for the following two weeks. You will also be contacted by text message to remind you to take your pills, to ask if you have taken your pills, and to send you a link to fill out questionnaires once daily. After the two weeks are over, you will again complete questionnaires and the online study session with tasks. Finally, two weeks after the second session, you will receive an email to fill out questionnaires online.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults 45-60

Exclusion Criteria: Following a structured telephone interview, participants with the following conditions will not be able to participate:

* certain active, uncontrolled medical disorders
* use of certain medications (e.g., hypnotic and psychotropic medication, steroid use, opioid use)
* psychiatric disorders (e.g., current major depression, bipolar disorder)

Other exclusion criteria may apply.

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2023-11-09 (Actual); Study Completion 2024-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi I Eisenberger, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Department of Psychology, Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naproxen | Placebo
Started | 65 | 79
Completed | 41 | 43
Not Completed | 24 | 36

BASELINE CHARACTERISTICS:
Population: Baseline includes those subjects who completed the study
Groups:
- Total: Total of all reporting groups
Arm/Group | Naproxen | Placebo | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 43 | 84
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (4.94) | 51.9 (5.11) | 51.9 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 60
  Male | 12 | 12 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity/Race: Asian | 4 | 3 | 7
  Ethnicity/Race: Black | 7 | 5 | 12
  Ethnicity/Race: Hispanic/Latino | 11 | 5 | 16
  Ethnicity/Race: Middle Eastern | 0 | 2 | 2
  Ethnicity/Race: White | 19 | 28 | 47
Region of Enrollment [Number; unit: participants]
  United States | 41 | 43 | 84

OUTCOME MEASURES:

1. Primary Outcome: Loneliness
Description: Changes in self-report measures of loneliness (University of California, Los Angeles (UCLA) Loneliness Scale) Scale ranges from 20-80 (though participants were included based on higher levels of loneliness, > 41). Higher values represent higher levels of loneliness.
Time Frame: T1: Baseline, T2: post-intervention (2 weeks later)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naproxen | Placebo
Number analyzed (Participants) | 41 | 43
score on a scale
  T1 Loneliness | 47.9 (10) | 46.9 (10.5)
  T2 Loneliness | 46.8 (9.43) | 44.6 (10.5)

2. Primary Outcome: Negative Picture Viewing Task
Description: Changes in ratings of negative pictures "To what extent is this picture positive or negative: from -5 (very negative) to +5 (very positive)" Lower scores indicate more negativity
Time Frame: T1: Baseline, T2: post-intervention (2 weeks later)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naproxen | Placebo
Number analyzed (Participants) | 41 | 43
score on a scale
  T1 Ratings of Pictures | -2.83 (1.58) | -2.60 (1.59)
  T2 Ratings of Pictures | -2.90 (1.61) | -2.66 (1.51)

3. Primary Outcome: Social Reward Task
Description: Changes in reaction time to close others vs. control image (measures in seconds) Faster reaction times indicate greater sensitivity; so lower scores (fewer seconds) indicate greater sensitivity to close others vs. control images
Time Frame: T1: Baseline, T2: post-intervention (2 weeks later)
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Naproxen | Placebo
Number analyzed (Participants) | 41 | 43
seconds
  T1 RT to close other vs. control | -0.012 (.056) | -.003 (.025)
  T2 RT to close other vs. control | -.020 (.112) | .002 (.054)

4. Secondary Outcome: Inflammatory Gene Expression
Description: Changes in inflammatory gene expression Values are the logged transformed values of a pre-specified composite of 19 representative proinflammatory genes (e.g., IL1B, IL6, COX2/PTGS2,TNF). Composite is in counts per million. Final scale is the logged value of this counts per million (logCPM). Higher numbers indicate greater inflammatory gene expression
Time Frame: T1: Baseline, T2: post-intervention (2 weeks later)
Measure: Mean (Standard Deviation); unit: logCPM
Arm/Group | Naproxen | Placebo
Number analyzed (Participants) | 41 | 43
logCPM
  T1 Inflammatory Composite | .070 (.352) | .057 (.357)
  T2 Inflammatory Composite | .042 (.292) | .001 (.345)

5. Secondary Outcome: Loneliness at Follow-up (2 Weeks Post-intervention)
Description: Changes in self-report measures of loneliness (University of California, Los Angeles (UCLA) Loneliness Scale) at follow-up, 2 weeks after the end of the intervention Scale ranges from 20-80 (though participants were included based on higher levels of loneliness, > 41). Higher values represent higher levels of loneliness.
Time Frame: T3: 2 weeks after the end of the intervention (4 weeks after the start of the intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naproxen | Placebo
Number analyzed (Participants) | 41 | 43
score on a scale | 45.1 (10.7) | 43.5 (10.8)

ADVERSE EVENTS:
Time Frame: Data were collected while participants were taking naproxen/placebo (2 weeks) as well as in the 2 weeks following the end of the intervention (T1 to T3).
Description: No adverse events
Arm/Group | Naproxen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/43
Other Adverse Events (participants affected / at risk) | 0/41 | 0/43

LIMITATIONS AND CAVEATS:
Because the study occurred during the COVID pandemic, we had to change our protocol to run all subjects online (drug/placebo was mailed to subjects as were blood collection devices). In addition, due to both budgetary issues and IRB concerns during the COVID pandemic, we had to shorten the planned intervention from 4 to 2 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-20): https://cdn.clinicaltrials.gov/large-docs/12/NCT03771612/Prot_SAP_000.pdf